CLINICAL TRIAL: NCT02768779
Title: IGHID 11601 - Measuring Antiretroviral Concentrations in Hair
Brief Title: ARV Concentrations in Hair
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-0398; R01AI122319-01 (NIH)
Record Dates: First submitted 2016-05-04; First posted 2016-05-11 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: HIV
Keywords: hair
MeSH Terms: interventions — Hair Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV negative and positive individuals: HIV Negative or HIV positive individuals, aged 18 years or older, who have been taking their ARV medication for at least 3 months and are adherent based on blood plasma HIV RNA of <50 copies/mL or HIV negative status. Hair analysis.
  Interventions: Other: Hair analysis

INTERVENTIONS:
Other: Hair analysis — Within the laboratory, experimental factors controlling IR-MALDESI response to key ARVs representing various drug classes will be systematically evaluated using the design of experiments (DOE) statistical approach (41,127) for an unbiased optimization of IRMALDESI response to each of the ARVs and their major metabolites. The goal will be to achieve a lower limit of quantification (LLOQ) below clinically relevant hair strand concentrations.

SUMMARY:
Hair samples from subjects on antiretroviral therapy, both HIV- and HIV+ patients with HIV RNA <50copies/mL for >6 months will be analyzed to investigate the influence of race, hair color and hair treatment on ARV response.

DETAILED DESCRIPTION:
A small thatch of hair (approximately 20 strands) will be collected from 85 participants who are currently taking antiretrovirals (ARVs). Hair collection will be evenly distributed into color cohorts: Black, Brown, Blonde and Grey. Participants will need to be >80% adherent to their medication and have had an undetectable HIV RNA VL within the previous 6 months. In the lab, samples will be used to develop IR-MALDESI MSI hair protocols for high sensitivity and accuracy to quantify ARVs in 5 therapeutic drug classes (Integrase Inhibitors, Nucleoside Reverse Transcriptase Inhibitors, Non-Nucleoside Reverse Transcriptase Inhibitors, Entry Inhibitors, Protease Inhibitors).

ELIGIBILITY:
Inclusion Criteria:

* HIV Negative or HIV positive individuals, aged 18 years or older, who have been taking their ARV medication for at least 3 months and are adherent based on blood plasma HIV RNA of <50 copies/mL or HIV negative status.

Exclusion Criteria:

* Subjects non-adherent to anti-retroviral regimen
* Subjects not willing or able to provide head hair sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hair samples will be collected from HIV negative and positive individuals taking ARVs.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
IR-MALDESI response to ARVs to be validated by LC-MS/MS analysis in hair before and after treatment with bleach | 1 year
  The effect of bleaching on hair collected from subjects adherence to an ARV regimen for >6 months
IR-MALDESI response to ARVs to be validated by LC-MS/MS analysis in hair before and after treatment with straighteners | 1 year
  The effect of straighteners on hair collected from subjects adherent to an ARV regimen for >6 months
IR-MALDESI response to ARVs to be validated by LC-MS/MS analysis in hair before and after treatment with hair color | 1 year
  The effect of hair color (dye) on hair collected from subjects adherent to an ARV regimen for >6 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamian MS, Golin CE, Shain LS, DeVellis B. Brief motivational interviewing to improve adherence to antiretroviral therapy: development and qualitative pilot assessment of an intervention. AIDS Patient Care STDS. 2004 Apr;18(4):229-38. doi: 10.1089/108729104323038900. PMID 15142353
- [Background] Adams JL, Patterson KB, Prince HM, Sykes C, Greener BN, Dumond JB, Kashuba AD. Single and multiple dose pharmacokinetics of dolutegravir in the genital tract of HIV-negative women. Antivir Ther. 2013;18(8):1005-13. doi: 10.3851/IMP2665. Epub 2013 Jul 31. PMID 23899439
- [Background] Adams JL, Sykes C, Menezes P, Prince HM, Patterson KB, Fransen K, Crucitti T, De Baetselier I, Van Damme L, Kashuba AD. Tenofovir diphosphate and emtricitabine triphosphate concentrations in blood cells compared with isolated peripheral blood mononuclear cells: a new measure of antiretroviral adherence? J Acquir Immune Defic Syndr. 2013 Mar 1;62(3):260-6. doi: 10.1097/QAI.0b013e3182794723. PMID 23111578
- [Background] Agius R, Kintz P; European Workplace Drug Testing Society. Guidelines for European workplace drug and alcohol testing in hair. Drug Test Anal. 2010 Aug;2(8):367-76. doi: 10.1002/dta.147. PMID 20818800
- [Background] Allen BC, Hack CE, Clewell HJ. Use of Markov Chain Monte Carlo analysis with a physiologically-based pharmacokinetic model of methylmercury to estimate exposures in US women of childbearing age. Risk Anal. 2007 Aug;27(4):947-59. doi: 10.1111/j.1539-6924.2007.00934.x. PMID 17958503
- [Background] Amico KR. Standard of Care for Antiretroviral Therapy Adherence and Retention in Care from the Perspective of Care Providers Attending the 5th International Conference on HIV Treatment Adherence. J Int Assoc Physicians AIDS Care (Chic). 2011 Sep-Oct;10(5):291-6. doi: 10.1177/1545109711406734. Epub 2011 May 10. PMID 21558490
- [Background] Amico KR, Fisher WA, Cornman DH, Shuper PA, Redding CG, Konkle-Parker DJ, Barta W, Fisher JD. Visual analog scale of ART adherence: association with 3-day self-report and adherence barriers. J Acquir Immune Defic Syndr. 2006 Aug 1;42(4):455-9. doi: 10.1097/01.qai.0000225020.73760.c2. PMID 16810111
- [Background] Amico KR, Mugavero M, Smith L, Crane H, Quinlivan E, Roytburd K, Golin CE, Zinski A, Modi R, Fredericksen R, Keruly J, Montue S. A brief provider survey to characterize retention and adherence standard of care support for patients in HIV care. 9th International Conference on HIV Treatment and Prevention Adherence, Miami FL, June 8-10, 2014.
- [Background] Appenzeller BM, Tsatsakis AM. Hair analysis for biomonitoring of environmental and occupational exposure to organic pollutants: state of the art, critical review and future needs. Toxicol Lett. 2012 Apr 25;210(2):119-40. doi: 10.1016/j.toxlet.2011.10.021. Epub 2011 Oct 31. PMID 22079616
- [Background] Arnold EA, Hazelton P, Lane T, Christopoulos KA, Galindo GR, Steward WT, Morin SF. A qualitative study of provider thoughts on implementing pre-exposure prophylaxis (PrEP) in clinical settings to prevent HIV infection. PLoS One. 2012;7(7):e40603. doi: 10.1371/journal.pone.0040603. Epub 2012 Jul 11. PMID 22792384
- See also: University of North Carolina website — http://www.unc.edu